CLINICAL TRIAL: NCT02475681
Title: A Randomized, Multicenter, Open-Label, 3 Arm Phase 3 Study of Obinutuzumab in Combination With Chlorambucil, Acalabrutinib (ACP-196) in Combination With Obinutuzumab, and Acalabrutinib Monotherapy in Subjects With Previously Untreated CLL
Brief Title: Acalabrutinib, Obinutuzumab and Chlorambucil in Treatment naïve CLL
Acronym: ElevateTN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACE-CL-007; 2023-509348-84-00 (Registry Identifier: CTIS (EU)); 2014-005582-73 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Results first posted 2023-01-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; obinutuzumab; Chlorambucil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A - Obinutuzumab in Combination with Chlorambucil (Active Comparator): Obinutuzumab IV infusions will be administered over a total of 6 treatment cycles starting at Cycle 1 Day 1. Chlorambucil will be orally administered on Days 1 and 15 of Cycles 1 through 6.
  Interventions: Drug: Obinutuzumab; Drug: Chlorambucil
- Arm B - Acalabrutinib in Combination with Obinutuzumab (Experimental): Obinutuzumab IV infusions will be administered over a total of 6 treatment cycles starting at Cycle 2 Day 1. Acalabrutinib (ACP-196) will be orally administered starting on Cycle 1 Day 1. Daily administration of Acalabrutinib (ACP-196) will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Drug: Obinutuzumab
- Arm C - Acalabrutinib Monotherapy (Experimental): Acalabrutinib (ACP-196) will be orally administered on Cycle 1 Day 1 until disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib
  Other Names: ACP-196 (Calquence)
  Arms: Arm B - Acalabrutinib in Combination with Obinutuzumab; Arm C - Acalabrutinib Monotherapy
Drug: Obinutuzumab
  Other Names: GAZYVA / GAZYVARO
  Arms: Arm A - Obinutuzumab in Combination with Chlorambucil; Arm B - Acalabrutinib in Combination with Obinutuzumab
Drug: Chlorambucil
  Other Names: LEUKERAN
  Arms: Arm A - Obinutuzumab in Combination with Chlorambucil

SUMMARY:
This Primary objective is evaluating the efficacy of obinutuzumab in combination with chlorambucil (Arm A) compared with acalabrutinib in combination with obinutuzumab (Arm B) for the treatment of previously untreated chronic lymphocytic leukemia (CLL). Secondary objectives: 1) To evaluate the efficacy of obinutuzumab in combination with chlorambucil (Arm A) versus acalabrutinib monotherapy (Arm C) based on IRC assessment of PFS per IWCLL 2008 criteria.

2)To compare obinutuzumab plus chlorambucil (Arm A) versus acalabrutinib plus obinutuzumab (Arm B) and obinutuzumab plus chlorambucil (Arm A) versus acalabrutinib monotherapy (Arm C) in terms of: IRC-assessed objective response rate (ORR); Tine to next treatment (TTNT); Overall Survival (OS)

DETAILED DESCRIPTION:
ELEVATE-TN is a global, phase 3, multicenter, open-label study in patients with treatment-naive chronic lymphocytic leukemia (CLL). Study enrollment is completed. The study randomized a total of 535 subjects in 142 study sites in 18 countries between 14 September 2015 through 08 February 2017. Patients were randomly assigned to receive Acalabrutinib and Obinutuzumab, Acalabrutinib monotherapy, or Obinutuzumab and oral Chlorambucil. The primary endpoint was progression-free survival between the two combination-therapy groups, defined as the time from randomization until disease progression by use of iwCLL 2008 criteria, or death, assessed by independent review committee (IRC). Crossover to Acalabrutinib was allowed in patients who progressed on Obinutuzumab-Chlorambucil.

The results of this study provide new evidence for therapy in patients with treatment-naive chronic lymphocytic leukemia by showing the efficacy of Acalabrutinib used with or without Obinutuzumab compared with chemoimmunotherapy.

Currently the study is in maintenance phase, with more than 430 subjects on study, to generate more evidence. We are not expecting any significant change in the near future.

ELIGIBILITY:
Inclusion Criteria

1. Men and women:

   a. ≥ 65 years of age OR b. > 18 and < 65 years of age, provided that they meet at least one of the following criteria: i. Creatinine clearance 30 to 69 mL/min using the Cockcroft-Gault equation ii. A score higher than 6 on the CIRS-G (Appendix L).
2. ECOG performance status of 0, 1, or 2.
3. Diagnosis of CD20+ CLL that meets published diagnostic criteria (Hallek 2008):

   1. Monoclonal B cells (either kappa or lambda light chain restricted) that are clonally co-expressing ≥ 1 B-cell marker (CD19, CD20, or CD23) and CD5.
   2. Prolymphocytes may comprise ≤ 55% of blood lymphocytes.
   3. Presence of ≥ 5 x 109 B lymphocytes/L (5000 μL) in the peripheral blood (at any point since diagnosis)
4. Active disease meeting ≥ 1 of the following IWCLL 2008 criteria for requiring treatment:

   1. Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia (hemoglobin < 10 g/dL) and/or thrombocytopenia (platelets < 100,000/μL).
   2. Massive (i.e., ≥ 6 cm below the left costal margin), progressive, or symptomatic splenomegaly.
   3. Massive nodes (i.e., ≥ 10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy.
   4. Progressive lymphocytosis with an increase of > 50% over a 2-month period or a LDT of < 6 months. LDT may be obtained by linear regression extrapolation of ALC obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In subjects with initial blood lymphocyte counts of < 30 x 109/L (30,000/μL), LDT should not be used as a single parameter to define indication for treatment. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL (e.g., infections) should be excluded.
   5. Autoimmune anemia and/or thrombocytopenia that is poorly responsive to standard therapy.
   6. Constitutional symptoms documented in the subject's chart with supportive objective measures, as appropriate, defined as ≥ 1 of the following disease-related symptoms or signs:

   i. Unintentional weight loss ≥ 10% within the previous 6 months before Screening.

   ii. Significant fatigue (i.e., ECOG performance status 2; inability to work or perform usual activities).

   iii. Fevers higher than 100.5°F or 38.0°C for 2 or more weeks before Screening without evidence of infection.

   iv. Night sweats for > 1 month before Screening without evidence of infection.
5. This criterion was deleted as of Protocol Amendment 3.
6. Meet the following laboratory parameters:

   1. ANC ≥ 750 cells/μL (0.75 x 109/L), or ≥ 500 cells/μL (0.50 x 109/L) in subjects with documented bone marrow involvement, and independent of growth factor support 7 days before assessment.
   2. Platelet count ≥ 50,000 cells/μL (50 x 109/L), or ≥ 30,000 cells/μL (30 x 109/L) in subjects with documented bone marrow involvement, and without transfusion support 7 days before assessment. Subjects with transfusion-dependent thrombocytopenia are excluded.
   3. Serum AST and ALT/SGPT ≤ 3.0 x ULN.
   4. Total bilirubin ≤ 1.5 x ULN.
   5. Estimated creatinine clearance (i.e., eGFR using Cockcroft-Gault) ≥ 30 mL/min
7. Able to receive all outpatient treatment, all laboratory monitoring, and all radiologic evaluations.
8. Women who are sexually active and can bear children must agree to use highly effective forms of contraception while on the study and for 2 days after the last dose of acalabrutinib or 18 months after the last dose of obinutuzumab in combination with chlorambucil, whichever is longer. Highly effective forms of contraception are defined in Section 6.4.4.
9. Men who are sexually active and can beget children must agree to use highly effective forms of contraception during the study and for 90 days after the last dose of obinutuzumab or chlorambucil, whichever is later. Highly effective forms of contraception are defined in Section 6.4.4.
10. Men must agree to refrain from sperm donation during the study and for 90 days after the last dose of obinutuzumab or chlorambucil, whichever is later.
11. Must be willing and able to adhere to the study visit schedule, understand and comply with other protocol requirements, and provide written informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations). Note vulnerable subjects, as defined in International Conference on Harmonisation (ICH) GCP, are not allowed on this protocol (e.g., prisoners or institutionalized subjects).

Exclusion Criteria:

1. Any prior systemic treatment for CLL (note: Prior localized radiotherapy is allowed).
2. Known CNS lymphoma or leukemia.
3. Known prolymphocytic leukemia or history of, or currently suspected, Richter's syndrome.
4. Missing or incomplete documentation of FISH results reflecting the presence or absence of 17p del and the percentage of cells with the deletion in subject records before randomization.
5. Uncontrolled AIHA or ITP defined as declining hemoglobin or platelet count secondary to autoimmune destruction within the screening period or requirement for high doses of steroids (> 20 mg daily of prednisone daily or equivalent).
6. Corticosteroid use > 20 mg within 1 week before first dose of study drug, except as indicated for other medical conditions such as inhaled steroid for asthma, topical steroid use, or as premedication for administration of study drug or contrast. For example, subjects requiring steroids at daily doses > 20 mg prednisone equivalent systemic exposure daily, or those who are administered steroids for leukemia control or WBC count lowering are excluded.
7. Major surgery within 4 weeks before first dose of study drug.
8. History of prior malignancy except for the following:

   1. Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years before Screening and felt to be at low risk for recurrence by treating physician.
   2. Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled non-melanomatous skin cancer.
   3. Adequately treated cervical carcinoma in situ without current evidence of disease.
9. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or QTc > 480 msec at screening.
10. Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or gastric bypass, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
11. Uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment) or ongoing intravenous anti-infective treatment.
12. Known history of infection with HIV. 13. Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.

14. Serologic status reflecting active hepatitis B or C infection. Subjects with hepatitis B core antibody positive who are surface antigen negative or who are hepatitis C antibody positive will need to have a negative PCR result before randomization. Those who are hepatitis B surface antigen positive or hepatitis B PCR positive and those who are hepatitis C PCR positive will be excluded.

15. History of stroke or intracranial hemorrhage within 6 months before randomization.

16. Known history of a bleeding diathesis (e.g., hemophilia, von Willebrand disease).

17. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days of first dose of study drug.

18. Requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole).

19. Breast feeding or pregnant. 20. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.

21. Concurrent participation in another therapeutic clinical trial. 22. Requires treatment with a strong CYP3A inhibitor/inducer. 23. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2025-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Clinical Study Information Center, Study Director — 1-877-240-9479 information.center@astrazeneca.com
Locations (143):
- United States (47):
  - Research Site, Goodyear, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Anaheim, California
  - Research Site, Los Angeles, California
  - Research Site, Oxnard, California
  - Research Site, Palo Alto, California
  - Research Site, Aurora, Colorado
  - Research Site, Lone Tree, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Niles, Illinois
  - Research Site, Lafayette, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, COL, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Billings, Montana
  - Research Site, Brick, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, Lake Success, New York
  - Research Site, New York, New York
  - Research Site, Blue Ash, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Sam Houston, Texas
  - Research Site, Houston, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Texas City, Texas
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Yakima, Washington
  - Research Site, Northwest WA, Wisconsin
- Australia (7):
  - Research Site, Darlinghurst
  - Research Site, Frankston
  - Research Site, Geelong
  - Research Site, South Brisbane
  - Research Site, Waratah NSW
  - Research Site, Wollongong
  - Research Site, Woodville
- Belgium (8):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Roeselare
  - Research Site, Wilrijk
  - Research Site, Yvoir
- Brazil (5):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Québec
  - Research Site, Saint John
  - Research Site, Winnipeg
- Chile (2):
  - Research Site, Santiago
  - Research Site, Temuco
- Colombia (2):
  - Research Site, Medellín
  - Research Site, Montería
- France (5):
  - Research Site, Bobigny
  - Research Site, Dijon
  - Research Site, Pierre-Bénite
  - Research Site, Strasbourg
  - Research Site, Villejuif
- Germany (5):
  - Research Site, Aschaffenburg
  - Research Site, Bielefeld
  - Research Site, Erlangen
  - Research Site, Heilbronn
  - Research Site, Warzburg
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kaposvár
  - Research Site, Szolnok
- Israel (10):
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Petah Tikvah
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
  - Research Site, Tiberias
- Italy (11):
  - Research Site, Alessandria
  - Research Site, Aviano
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Parma
  - Research Site, Ravenna
  - Research Site, Rimini
  - Research Site, Rome
  - Research Site, Rozzano
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Otahuhu
  - Research Site, Tauranga
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Słupsk
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Santander
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Örebro
- United Kingdom (9):
  - Research Site, Bournemouth
  - Research Site, Cambridge
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Plymouth
  - Research Site, Southampton
  - Research Site, Truro
  - Research Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Sharman JP, Egyed M, Jurczak W, Skarbnik A, Patel K, Flinn IW, Kamdar M, Munir T, Walewska R, Hughes M, Fogliatto LM, Herishanu Y, Banerji V, Follows G, Walker P, Ghia P, Janssens A, Byrd JC, Ferrant E, Ferrajoli A, Wierda WG, Wachira CW, Suterwala BT, Miranda P, Munugalavadla V, Wun CC, Woyach JA. Acalabrutinib-obinutuzumab improves survival vs chemoimmunotherapy in treatment-naive CLL in the 6-year follow-up of ELEVATE-TN. Blood. 2025 Sep 11;146(11):1276-1285. doi: 10.1182/blood.2024024476. PMID 40198878
- [Derived] Kittai AS, Allan JN, James D, Bridge H, Miranda M, Yong ASM, Fam F, Roos J, Shetty V, Skarbnik A, Davids MS. An indirect comparison of acalabrutinib with and without obinutuzumab vs zanubrutinib in treatment-naive CLL. Blood Adv. 2024 Jun 11;8(11):2861-2869. doi: 10.1182/bloodadvances.2023012142. PMID 38598745
- [Derived] Sharman JP, Egyed M, Jurczak W, Skarbnik A, Pagel JM, Flinn IW, Kamdar M, Munir T, Walewska R, Corbett G, Fogliatto LM, Herishanu Y, Banerji V, Coutre S, Follows G, Walker P, Karlsson K, Ghia P, Janssens A, Cymbalista F, Woyach JA, Salles G, Wierda WG, Izumi R, Munugalavadla V, Patel P, Wang MH, Wong S, Byrd JC. Acalabrutinib with or without obinutuzumab versus chlorambucil and obinutuzmab for treatment-naive chronic lymphocytic leukaemia (ELEVATE TN): a randomised, controlled, phase 3 trial. Lancet. 2020 Apr 18;395(10232):1278-1291. doi: 10.1016/S0140-6736(20)30262-2. PMID 32305093
- See also: Statistical Analysis Plan Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-007&attachmentIdentifier=8ef87193-534b-4eea-8fb3-3f20652f1c3e&fileName=ace-cl-007-statistical-analysis-plan-redact.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-007&attachmentIdentifier=8cdfe1aa-e61b-4f7a-8624-2f1bc0df4f3b&fileName=ace-cl-007-protocol-redact.pdf&versionIdentifier=
- See also: Redacted Clinical Study Report synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-007&attachmentIdentifier=33003026-e482-482b-a4ee-845f714960e3&fileName=ace-cl-007-clinical-study-report-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, multicenter, open-label, 3 arm phase 3 study of Obinutuzumab in combination with Chlorambucil (Chlb+Obin), Acalabrutinib in combination with Obinutuzumab (Acala+Obin), and Acalabrutinib monotherapy (Acala) in subjects with previously untreated chronic lymphocytic leukemia. A total of 535 subjects recruited from 142 sites in 18 countries were randomized (1:1:1) as follows: 179/179 /177 subjects in Acla+Obin arm / Acala arm / Chlb+Obin arm respectively.
Groups:
- Arm A: Obinutuzumab in Combination With Chlorambucil: Obinutuzumab IV infusions will be administered over a total of 6 treatment cycles, starting from cycle1 to cycle 6. Chlorambucil will be orally administered on Days 1 and 15 of Cycles 1 through 6. At investigator discretion, subjects randomized to this treatment arm, who had IRC-confirmed disease progression, were eligible to receive crossover treatment with single-agent acalabrutinib at 100 mg BID until disease progression or unacceptable toxicity.
- Arm B: Acalabrutinib in Combination With Obinutuzumab: Acalabrutinib (ACP-196) will be orally administered starting on Cycle 1 Day 1. Obinutuzumab IV infusions will be administered over a total of 6 treatment cycles, starting in Cycle 2 Day 1. Daily administration of Acalabrutinib (ACP-196) will continue until disease progression or unacceptable toxicity.
- Arm C: Acalabrutinib Monotherapy: Acalabrutinib (ACP-196) will be orally administered on Cycle 1 Day 1 until disease progression or unacceptable toxicity. Acalabrutinib
Period: Overall Study
Arm/Group | Arm A: Obinutuzumab in Combination With Chlorambucil | Arm B: Acalabrutinib in Combination With Obinutuzumab | Arm C: Acalabrutinib Monotherapy
Started (Randomized) | 177 | 179 | 179
Crossed Over From Arm A to Arm C | 45 | 0 | 0
Completed | 145 | 0 | 0
Not Completed | 32 | 179 | 179
Not completed — Death | 16 | 6 | 9
Not completed — Physician Decision | 0 | 3 | 1
Not completed — Withdrawal by Subject | 12 | 6 | 9
Not completed — Lost to Follow-up | 2 | 1 | 3
Not completed — Ongoing in Study | 0 | 163 | 157
Not completed — Reasons other than above listed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat (ITT) population, which included all randomized participants grouped according to assigned treatment.
Groups:
- Obinutuzumab in Combination With Chlorambucil: Obinutuzumab IV infusions will be administered over a total of 6 treatment cycles starting at Cycle 1 Day 1. Chlorambucil will be orally administered on Days 1 and 15 of Cycles 1 through 6. Obinutuzumab Chlorambucil
- Acalabrutinib in Combination With Obinutuzumab: Obinutuzumab IV infusions will be administered over a total of 6 treatment cycles starting at Cycle 2 Day 1. Acalabrutinib (ACP-196) will be orally administered starting on Cycle 1 Day 1. Daily administration of Acalabrutinib (ACP-196) will continue until disease progression or unacceptable toxicity. Acalabrutinib Obinutuzumab
- Acalabrutinib Monotherapy: Acalabrutinib will be orally administered on Cycle 1 Day 1 until disease progression or unacceptable toxicity. Acalabrutinib
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab in Combination With Chlorambucil | Acalabrutinib in Combination With Obinutuzumab | Acalabrutinib Monotherapy | Total
Number analyzed (Participants) | 177 | 179 | 179 | 535
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 35 | 28 | 87
  >=65 years | 153 | 144 | 151 | 448
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 68 | 68 | 207
  Male | 106 | 111 | 111 | 328
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 2 | 11 | 24
  Not Hispanic or Latino | 156 | 169 | 156 | 481
  Unknown or Not Reported | 10 | 8 | 12 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 4 | 5 | 4 | 13
  White | 165 | 164 | 170 | 499
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 5 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 5 | 5 | 3 | 13
  France | 3 | 3 | 1 | 7
  Germany | 3 | 1 | 3 | 7
  Italy | 11 | 9 | 5 | 25
  Spain | 7 | 3 | 3 | 13
  Sweden | 1 | 3 | 3 | 7
  United Kingdom | 12 | 16 | 17 | 45
  Brazil | 4 | 5 | 5 | 14
  Chile | 2 | 0 | 3 | 5
  Colombia | 1 | 0 | 0 | 1
  Canada | 7 | 8 | 7 | 22
  United States | 54 | 56 | 63 | 173
  Hungary | 17 | 26 | 15 | 58
  Lithuania | 9 | 2 | 6 | 17
  Poland | 14 | 20 | 25 | 59
  Australia | 9 | 9 | 8 | 26
  New Zealand | 8 | 4 | 5 | 17
  Israel | 10 | 9 | 7 | 26
IXRS Randomization Stratification Factor: Presence of 17p Deletion [Count of Participants; unit: Participants]
  Yes | 17 | 21 | 19 | 57
  No | 160 | 158 | 160 | 478
IXRS Randomization Stratification Factor: ECOG Performance Status [Count of Participants; unit: Participants] — Lower Grade is Better. 0=Fully active; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all selfcare but unable to carry out any work activities;
  Participants
    0-1 (0=Fully Active; 1 =Restricted in Physically Strenuous Activity) | 168 | 169 | 167 | 504
    2 (2=Ambulatory and capable of all selfcare but unable to carry out any work activities) | 9 | 10 | 12 | 31
IXRS Randomization Stratification Factor: Geographic Region [Count of Participants; unit: Participants]
  North America and West Europe | 103 | 104 | 105 | 312
  Other | 74 | 75 | 74 | 223

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival by IRC (Independent Review Committee) Assessment in Arm A Compared to Arm B
Description: To evaluate the efficacy of obinutuzumab in combination with chlorambucil (Arm A) compared with acalabrutinib in combination with obinutuzumab (Arm B) based on IRC assessment of progression-free survival (PFS) per International Workshop on Chronic Lymphocytic Leukemia criteria (IWCLL; Hallek et al. 2008) with incorporation of the clarification for treatment-related lymphocytosis (Cheson et al. 2012), hereafter referred to as IWCLL 2008 criteria, in subjects with previously untreated CLL. PFS, defined as the time from date of randomization to the date of first IRC-assessed disease progression or death due to any cause, whichever comes first.
Time Frame: IRC assessments were done from randomization date until disease progression or death or IRC discontinuation date on 08Feb2019 (as the IA based on this data cutoff date showed the study crossing superiority boundary) whichever comes first up to 40 months.
Population: Intent to Treat (ITT)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Obinutuzumab in Combination With Chlorambucil | Arm B: Acalabrutinib in Combination With Obinutuzumab
Number analyzed (Participants) | 177 | 179
Months | 22.6 [20.2 to 27.8] | NA [NA to NA] — Median and 95% CIs for Arm B = NA (not reached) since insufficient numbers of subjects with events (Range = 0.0+ to 39.4+ months). "+" indicates a value from a censored subject.
Statistical Analysis 1: Comparison: Arm A: Obinutuzumab in Combination With Chlorambucil vs Arm B: Acalabrutinib in Combination With Obinutuzumab; The primary test to compare PFS between treatment arms was the two-sided log-rank test, stratified by randomization stratification factors. The estimate of the HR (Arm B/Arm A) and the corresponding 95% CI was computed using a Cox proportional hazards model stratified by randomization stratification factors. Randomization stratification factors were based on the data recorded in IXRS; Test type: Superiority; p < 0.0001, Log Rank; Stratified by randomization stratification factors as recorded in IXRS; Hazard Ratio (HR) = 0.1, 95% CI 2-sided [0.06 to 0.17]

2. Secondary Outcome: Progression-free Survival by IRC Assessment Arm A Versus Arm C
Description: To evaluate the efficacy of obinutuzumab in combination with chlorambucil (Arm A) compared with acalabrutinib monotherapy (Arm C) based on IRC assessment of progression-free survival (PFS) per International Workshop on Chronic Lymphocytic Leukemia criteria (IWCLL; Hallek et al. 2008) with incorporation of the clarification for treatment-related lymphocytosis (Cheson et al. 2012), hereafter referred to as IWCLL 2008 criteria, in subjects with previously untreated CLL. PFS, defined as the time from date of randomization to the date of first IRC-assessed disease progression or death due to any cause, whichever comes first.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Obinutuzumab in Combination With Chlorambucil | Arm C: Acalabrutinib Monotherapy
Number analyzed (Participants) | 177 | 179
Months | 22.6 [20.2 to 27.6] | NA [34.2 to NA] — The median PFS for Arm C was not reached (Range = 0.0+ to 39.5+ months). "+" indicates a value from a censored subject.
Statistical Analysis 1: Comparison: Arm A: Obinutuzumab in Combination With Chlorambucil vs Arm C: Acalabrutinib Monotherapy; The test to compare PFS between treatment Arms A and C was the two-sided log-rank test, stratified by randomization stratification factors. The estimate of the HR and the corresponding 95% CI was computed using a Cox proportional hazards model stratified by randomization stratification factors. Randomization stratification factors were based on the data recorded in IXRS; Test type: Superiority; p < 0.0001, Log Rank; Stratified by randomization stratification factors as recorded in IXRS; Hazard Ratio (HR) = 0.2, 95% CI 2-sided [0.13 to 0.30]

3. Secondary Outcome: IRC-assessed Objective Response Rate (ORR) in Arm A Versus Arm B and Arm A Versus Arm C
Description: ORR was defined as the proportion of subjects who achieved a best response of CR, CRi, nPR, or PR at or before initiation of subsequent anticancer therapy. ORR including PRL was defined as the proportion of subjects who achieved a best response of CR, CRi, nPR, PR or PRL at or before initiation of subsequent anticancer therapy
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Obinutuzumab in Combination With Chlorambucil | Arm B: Acalabrutinib in Combination With Obinutuzumab | Arm C: Acalabrutinib Monotherapy
Number analyzed (Participants) | 177 | 179 | 179
percentage of participants | 78.5 [71.9 to 83.9] | 93.9 [89.3 to 96.5] | 85.5 [79.6 to 89.9]
Statistical Analysis 1: Comparison: Arm A: Obinutuzumab in Combination With Chlorambucil vs Arm B: Acalabrutinib in Combination With Obinutuzumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenzel test with adjustment for randomization stratification factors as recorded in IXRS; Risk Difference (RD) = 15.3, 95% CI 2-sided [8.3 to 22.3]
Statistical Analysis 2: Comparison: Arm A: Obinutuzumab in Combination With Chlorambucil vs Arm C: Acalabrutinib Monotherapy; Test type: Superiority; p = 0.0763, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenzel test with adjustment for randomization stratification factors as recorded in IXRS; Risk Difference (RD) = 6.9, 95% CI 2-sided [-1.0 to 14.9]

4. Secondary Outcome: Time to Next Treatment (TTNT) in Arm A Versus Arm B and Arm A Versus Arm C
Description: TTNT was defined as the time from randomization to start date of non-protocol specified subsequent anticancer therapy for CLL or death due to any cause, whichever came first. TTNT was analyzed in the same fashion as that for the primary efficacy analysis
Time Frame: From randomization date to start of non-protocol specified subsequent anticancer therapy for CLL or death due to any cause, whichever came first assessed up to 40 months of follow-up.
Population: Intent to Treat (ITT)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Obinutuzumab in Combination With Chlorambucil | Arm B: Acalabrutinib in Combination With Obinutuzumab | Arm C: Acalabrutinib Monotherapy
Number analyzed (Participants) | 177 | 179 | 179
Months | NA [28.9 to NA] — The median TTNT was not reached for obinutuzumab+chlorambucil (range: 0.0+ to 39.6+ months). "+" indicates a value from a censored subject. | NA [NA to NA] — The median TTNT was not reached for acalabrutinib+obinutuzumab (range: 1.3-40.3+ months). "+" indicates a value from a censored subject. | NA [NA to NA] — The median TTNT was not reached for acalabrutinib monotherapy (range: 0.1+ to 40.1+ months). "+" indicates a value from a censored subject.
Statistical Analysis 1: Comparison: Arm A: Obinutuzumab in Combination With Chlorambucil vs Arm B: Acalabrutinib in Combination With Obinutuzumab; The test to compare TTNT between treatment Arms A versus B and Arms A versus C was the two-sided log-rank test, stratified by randomization stratification factors. The estimate of the HR and the corresponding 95% CI was computed using a Cox proportional hazards model stratified by randomization stratification factors. Randomization stratification factors were based on the data recorded in IXRS; Test type: Superiority; p < 0.0001, Log Rank; Stratified by randomization stratification factors as recorded in IXRS; Hazard Ratio (HR) = 0.14, 95% CI 2-sided [0.08 to 0.26]
Statistical Analysis 2: Comparison: Arm A: Obinutuzumab in Combination With Chlorambucil vs Arm C: Acalabrutinib Monotherapy; Test type: Superiority; p < 0.0001, Log Rank — P-value based on stratified by randomization stratification factors as recorded in IXRS; Stratified by randomization stratification factors as recorded in IXRS; Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.15 to 0.40]

5. Secondary Outcome: Overall Survival (OS) in Arm A Versus Arm B and Arm A Versus Arm C
Description: OS was defined as the time from the date of randomization to death due to any cause.
Time Frame: From randomization date until death, withdrawal by subject, lost to follow-up, or by analysis data cut off date on 08Feb2019 whichever comes first up to 40 months of follow-up.
Population: Intent to Treat (ITT)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Obinutuzumab in Combination With Chlorambucil | Arm B: Acalabrutinib in Combination With Obinutuzumab | Arm C: Acalabrutinib Monotherapy
Number analyzed (Participants) | 177 | 179 | 179
Months | NA [NA to NA] — The median and corresponding 95% CI for the OS in Arm A was not reached due to insufficient subjects with events (Range of OS =1.7 to 40.4+ months). "+" indicates a value from a censored subject. | NA [NA to NA] — The median and corresponding 95% CI for the OS in Arm B was not reached due to insufficient subjects with events (Range of OS =0.1+ to 40.8+ months). "+" indicates a value from a censored subject. | NA [NA to NA] — The median and corresponding 95% CI for the OS in Arm C was not reached due to insufficient subjects with events. (Range of OS = 0.0+ to 40.7+ months) "+" indicates a value from a censored subject.
Statistical Analysis 1: Comparison: Arm A: Obinutuzumab in Combination With Chlorambucil vs Arm B: Acalabrutinib in Combination With Obinutuzumab; The test to compare overall survival between treatment Arms A versus B and Arms A versus C was the two-sided log-rank test, stratified by randomization stratification factors. The estimate of the HR and the corresponding 95% CI was computed using a Cox proportional hazards model stratified by randomization stratification factors. Randomization stratification factors were based on the data recorded in IXRS; Test type: Superiority; p = 0.0577, Log Rank; Stratified by randomization stratification factors as recorded in IXRS; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.21 to 1.06]
Statistical Analysis 2: Comparison: Arm A: Obinutuzumab in Combination With Chlorambucil vs Arm C: Acalabrutinib Monotherapy; Test type: Superiority; p = 0.1556, Log Rank; Stratified by randomization stratification factors as recorded in IXRS; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.28 to 1.27]

ADVERSE EVENTS:
Time Frame: All adverse events were reported from randomization date until 30 days after the last dose of study drug or the start of new anticancer therapy (whichever comes first) up to 61 months. After this period, investigators reported SAEs or other AEs of concern that are believed to be related to prior treatment with study drug up to 5 years.
Description: Data presented under All-Cause Mortality table are based on ITT Population (all randomized) as those presented in Participant Flow. Data presented under SAE and AE Tables are based on Safety Population (Subjects received at least one dose of study drug).
Groups:
- Arm C: Acalabrutinib Monotherapy: Acalabrutinib will be orally administered on Cycle 1 Day 1 until disease progression or unacceptable toxicity. Acalabrutinib
- Arm A Cross-over: Obinutuzumab+Chlorambucil Crossover to Acalabrutinib Monotherapy: Obinutuzumab + Chlorambucil Crossover to Acalabrutinib 100 mg twice daily monotherapy
Arm/Group | Arm A: Obinutuzumab in Combination With Chlorambucil | Arm B: Acalabrutinib in Combination With Obinutuzumab | Arm C: Acalabrutinib Monotherapy | Arm A Cross-over: Obinutuzumab+Chlorambucil Crossover to Acalabrutinib Monotherapy
All-Cause Mortality (participants affected / at risk) | 17/177 | 9/179 | 11/179 | 2/45
Serious Adverse Events (participants affected / at risk) | 37/169 | 69/178 | 57/179 | 6/45
Other Adverse Events (participants affected / at risk) | 167/169 | 171/178 | 170/179 | 37/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Obinutuzumab in Combination With Chlorambucil (N=169) | Arm B: Acalabrutinib in Combination With Obinutuzumab (N=178) | Arm C: Acalabrutinib Monotherapy (N=179) | Arm A Cross-over: Obinutuzumab+Chlorambucil Crossover to Acalabrutinib Monotherapy (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 3 | 2 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 3 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 1 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 2 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 12 | 5 | 0
Urosepsis (Infections and infestations) | 0 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 2 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 3 | 0
Bacterial sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Vascular access site infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Dacryocystitis (Infections and infestations) | 1 | 0 | 0 | 0
Disseminated cryptococcosis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 4 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Costal cartilage fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Pseudohyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 8 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Obinutuzumab in Combination With Chlorambucil (N=169) | Arm B: Acalabrutinib in Combination With Obinutuzumab (N=178) | Arm C: Acalabrutinib Monotherapy (N=179) | Arm A Cross-over: Obinutuzumab+Chlorambucil Crossover to Acalabrutinib Monotherapy (N=45)
Neutropenia (Blood and lymphatic system disorders) | 76 | 56 | 19 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 23 | 13 | 3
Anaemia (Blood and lymphatic system disorders) | 20 | 21 | 25 | 0
Diarrhoea (Gastrointestinal disorders) | 36 | 69 | 62 | 8
Nausea (Gastrointestinal disorders) | 53 | 36 | 40 | 9
Constipation (Gastrointestinal disorders) | 17 | 25 | 20 | 5
Vomiting (Gastrointestinal disorders) | 19 | 24 | 22 | 2
Abdominal pain (Gastrointestinal disorders) | 12 | 11 | 9 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 11 | 8 | 1
Dyspepsia (Gastrointestinal disorders) | 8 | 9 | 14 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 3 | 11 | 2
Fatigue (General disorders) | 29 | 50 | 33 | 6
Pyrexia (General disorders) | 35 | 23 | 12 | 5
Oedema peripheral (General disorders) | 12 | 22 | 16 | 3
Chills (General disorders) | 14 | 20 | 8 | 0
Asthenia (General disorders) | 10 | 17 | 9 | 1
Peripheral swelling (General disorders) | 4 | 9 | 9 | 2
Influenza like illness (General disorders) | 4 | 8 | 12 | 1
Upper respiratory tract infection (Infections and infestations) | 14 | 38 | 33 | 6
Urinary tract infection (Infections and infestations) | 8 | 22 | 22 | 3
Nasopharyngitis (Infections and infestations) | 7 | 20 | 17 | 4
Sinusitis (Infections and infestations) | 6 | 16 | 12 | 0
Bronchitis (Infections and infestations) | 5 | 15 | 14 | 2
Pneumonia (Infections and infestations) | 5 | 19 | 13 | 1
Herpes zoster (Infections and infestations) | 4 | 11 | 5 | 1
Contusion (Injury, poisoning and procedural complications) | 7 | 42 | 27 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 67 | 24 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 14 | 11 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 18 | 10 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 12 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 9 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 8 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 39 | 28 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 25 | 25 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 22 | 11 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 14 | 15 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 13 | 10 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 9 | 10 | 1
Headache (Nervous system disorders) | 20 | 71 | 66 | 10
Dizziness (Nervous system disorders) | 10 | 32 | 21 | 4
Paraesthesia (Nervous system disorders) | 4 | 10 | 5 | 0
Insomnia (Psychiatric disorders) | 16 | 16 | 15 | 3
Anxiety (Psychiatric disorders) | 5 | 9 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 39 | 33 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 15 | 12 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 13 | 10 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 13 | 8 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 12 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 21 | 25 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 14 | 16 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 11 | 15 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 7 | 9 | 0
Hypotension (Vascular disorders) | 5 | 14 | 6 | 1
Hypertension (Vascular disorders) | 6 | 11 | 8 | 1
Haematoma (Vascular disorders) | 1 | 9 | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator will not publish or publicly present any study results without prior approval or prior to 12 months following completion of the study.

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT02475681/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT02475681/SAP_001.pdf